CLINICAL TRIAL: NCT04170894
Title: Radiofrequency Ablation of Atrial Fibrillation Under Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Northwell Health (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-04020216
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Radiofrequency Ablation; Ablation; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apnea (Experimental): Patients will undergo an atrial fibrillation ablation and will have induced periods of apnea throughout the procedure.
  Interventions: Other: Periods of Apnea
- Control (Active Comparator): Patients who choose not to participate in the apnea arm will have the opportunity to consent to the control arm. These patients will undergo an atrial fibrillation ablation per standard of care without periods of apnea throughout the procedure. This data will be collected to use as a comparator to the apnea arm.
  Interventions: Other: Control Arm - No Periods of Apnea

INTERVENTIONS:
Other: Periods of Apnea — Periods of apnea throughout atrial fibrillation ablation.
  Arms: Apnea
Other: Control Arm - No Periods of Apnea — Standard of care atrial fibrillation ablation.
  Arms: Control

SUMMARY:
This study seeks to assess the effect of apnea (breath hold) during atrial fibrillation (AF) ablation by having all ablations performed under apnea. By prospectively studying the effects of apnea on AF ablation, the investigators wish to demonstrate its feasibility, safety and impact on patient outcomes. This is a prospective study that includes both an apnea arm and a control arm. The subjects who consent to the apnea arm will undergo an atrial fibrillation ablation with periods of apnea. The subjects who consent to the control arm will agree to have their data from their standard of care atrial fibrillation be collected for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years old.
* Symptomatic paroxysmal atrial fibrillation.

Exclusion Criteria:

* Patients with persistent or permanent atrial fibrillation or prior atrial fibrillation ablation.
* Significant chronic obstructive pulmonary disease (such as those requiring home oxygen).
* Severe pulmonary hypertension.
* Other intrinsic lung pathology such as interstitial lung disease.
* Severe systolic dysfunction defined as left ventricular ejection fraction < 30%.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Catheter Stability Metrics as measured by contact force variability. | Day 1
  Contact force variability: Catheter stability metrics will be calculated as standard deviations of contact forces measured during the course of reach ablation region. Contact forces and their standard deviations will range between 0 and 60 grams.
Catheter Stability Metrics as measured by maximum and minimum contact force. | Day 1
  Maximum contact force: range between 0 and 60 grams
Catheter Stability Metrics as measured by average contact force. | Day 1
  Average contact force: range between 0 and 60 grams
Catheter Stability Metrics as measured by catheter displacement. | Day 1
  Catheter displacement (mean): range 0-10 mm
Efficacy as measured by time to pulmonary vein isolation. | Day 1
  Time to pulmonary vein isolation (minutes): expected range 60 - 180 minutes
Efficacy as measured by percentage of veins isolated after first pass. | Day 1
  Percentage of veins isolated after first pass: 0-100%
Catheter Stability Metrics as measured by time to impedance drop. | Day 1
  Time to 5 ohm and 10 ohm impedance drop: range 1 to 60 seconds

SECONDARY OUTCOMES:
Procedural time as measured by the length of time from start to end of procedure. | Day 1
  Length of procedure time determined by time lapsed per report from start of procedure to end of procedure.
Clinical Outcomes as measured by recurrence of atrial fibrillation at six months post procedure. | month six
  Percentage of subjects with atrial fibrillation on 5 day event monitor at 6 months post-intervention.
Clinical Outcomes as measured by recurrence of atrial fibrillation at 12 months post procedure. | month 12
  Percentage of subjects with atrial fibrillation on 5 day event monitor at 12 months post-intervention.
Safety, as measured by number of subjects with at least one adverse event. | End of study (12 months)
  Adverse events will include any unfavorable and unintended sign, symptom, or disease temporally associated with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jim Cheung, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (6):
- United States (6):
  - Southside Hospital, Bay Shore, New York
  - North Shore Hospital, Manhasset, New York
  - New York Presbyterian Hospital - Weill Cornell Medicine, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Long Island Jewish Medical Center, Queens, New York
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gabriels JK, Ying X, Purkayastha S, Braunstein E, Liu CF, Markowitz SM, Mountantonakis S, Thomas G, Goldner B, Willner J, Goyal R, Ip JE, Lerman BB, Carter J, Bereanda N, Fitzgerald MM, Anca D, Patel A, Cheung JW. Safety and Efficacy of a Novel Approach to Pulmonary Vein Isolation Using Prolonged Apneic Oxygenation. JACC Clin Electrophysiol. 2023 Apr;9(4):497-507. doi: 10.1016/j.jacep.2022.10.030. Epub 2023 Jan 18. PMID 36752460